CLINICAL TRIAL: NCT05619107
Title: Transauricular Nerve Stimulation to Enhance Exercise Capacity: Protocol for a Double-blind, Open Crossover, Randomised Sham-controlled Trial
Brief Title: Boosting Exercise cApaCity With autOnomic Neuromodulation
Acronym: BEACON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 299987
Record Dates: First submitted 2022-10-18; First posted 2022-11-16 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2022-10

CONDITIONS: Aging; Inflammation; Cardiovascular Diseases
Keywords: Neuromodulation; Exercise Training
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Double-blind, open crossover, randomised sham-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and investigators are blinded to treatment allocations throughout data collection and analysis. Participants and investigators are also masked to the outcomes data, which will be analysed offline by an independent trial statistician not involved with patient recruitment/device application who is masked to the treatment allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transauricular nerve stimulation (Active Comparator): Using a training device, two conductive clips are placed securely on both the left and right tragus areas of the outer ear. Using parameters we have identified through systematic review, electrical stimulation (pulse width:200μs; frequency:30Hz) is initiated at 10mA, until the participant feels a 'tingling' sensation within 20s of commencing. At this point the current is reduced to a level just below this perceptible threshold (20-60 mA), which is defined as the 'prescription dose'. The participant then receives another active device set at the 'prescription dose'.
  Interventions: Device: Active Transauricular nerve stimulation
- Sham transauricular nerve stimulation (Sham Comparator): Using a training device, two conductive clips are placed securely on both the left and right tragus areas of the outer ear. Using parameters we have identified through systematic review, electrical stimulation (pulse width:200μs; frequency:30Hz) is initiated at 10mA, until the participant feels a 'tingling' sensation within 20s of commencing (Figure 2). At this point the current is reduced to a level just below this perceptible threshold (20-60 mA), which is defined as the 'prescription dose'. The participant then receives another device set at the 'prescription dose' but this sham device is disabled from delivering any current .
  Interventions: Device: Sham transauricular nerve stimulation

INTERVENTIONS:
Device: Active Transauricular nerve stimulation — The first allocated intervention will be undertaken for 30 minutes. The electrode placement and stimulation parameters are described in the arm/group section. After the 30-minute intervention, day 1 of the protocol will be complete. The investigator will remain present in the room with the participant to ensure compliance and adherence to the protocol. The allocated intervention will then be repeated by the participant at a similar time of day for 7 consecutive days. The investigator will arrange video-calls with the participant whilst off-site to ensure ongoing compliance and adherence to the protocol. On the seventh day, participants return to the clinical research facility to take the final first allocated intervention. A 14-day rest period will follow. Then the participants will perform the same 7-day protocol for the opposite intervention to their first treatment allocation.
  Arms: Active transauricular nerve stimulation
Device: Sham transauricular nerve stimulation — Protocol as for active but sham ear leads are applied, unable to deliver current.
  Arms: Sham transauricular nerve stimulation

SUMMARY:
Background: Exercise performance is a key predictor for healthy ageing. Laboratory and clinical data have shown strength of a nerve called the vagus nerve, which is lost during age-related disease processes, determines exercise performance. The investigators describe a study protocol designed to test the hypothesis that stimulation of the ear (where the vagus nerve can be safely stimulated) may improve exercise performance alongside beneficial changes in vagus nerve activity in human volunteers.

Methods. 28 healthy participants aged 18-75y will be randomly allocated to electrical ear stimulation or placebo treatment for 30 minutes at the same time of day, for 7 consecutive days. Heart monitoring, exercise bike testing, a simple sit-to-stand test and blood sampling will be performed immediately before the first day's intervention and after the last day's intervention. Participants and investigators will be masked to the treatment allocations and analyses. After a 14-day break, participants will perform the same protocol for the opposite intervention to their first treatment allocation. The primary outcome will be the change in VO2Peak (the best measure of exercise performance) following stimulation or placebo protocol. Secondary outcomes include reduction in heart rate after ending the exercise bike test, reduction from peak heart rate after standing from sitting, beat-to-beat heart rate measures and blood inflammatory marker levels. These outcomes will measure exercise performance and vagus nerve function. Safety and complications of the intervention will also be recorded. The study was approved by the NHS Research Ethics Committee (21/LO/0856).

Discussion. This 'first-in-man' study will explore whether non-invasive vagus nerve stimulation safely boosts exercise performance and/or vagus nerve activity using electrical ear stimulation, providing data for a device-based approach that may be broadly generalisable to improving health outcomes.

DETAILED DESCRIPTION:
Background A cardinal feature of acute tissue injury/systemic inflammation is the development of autonomic dysfunction, characterised by sustained sympathetic hyperactivity and loss of vagal function. Elevated resting heart rate is repeatedly associated with both cardiovascular morbidity and all-cause mortality in the general population. Vagal tone, which declines variably during ageing processes, is the chief determinant of resting heart rate. Healthy ageing is characterised by lower sympathetic and preserved vagal activity, reflected by lower resting heart rate. The gold-standard measure of vagal tone is heart rate recovery (HRR), obtainable from exercise testing. Loss of vagal tone in humans - as quantified by HRR - is associated with lower peak aerobic exercise capacity, a major barrier to rehabilitation. Persistent sympathetic hyperactivity downregulates G-protein coupled β-receptor recycling. This impairs cardiac function, lowers exercise capacity and increases systemic inflammation, thereby promoting cardiometabolic disease. Exercise tolerance may be enhanced by dedicated exercise training programmes, even in healthy individuals. Greater exercise capacity is linked with lower risks of cardiovascular disease, Type 2 diabetes, malignancy, osteoporosis, depression and premature death.

Although in healthy ageing cardiac vagal tone is predominantly determined by genetic factors, with strong associations identified between HRR and various genes expressed by key autonomic pathway components, vagal neuromodulation techniques have gained traction. Laboratory and clinical translational data have shown restoring (or preventing the loss of) vagal activity may therefore offer a therapeutic target to help optimise cardiopulmonary fitness and improve health outcomes. Stimulation of the dorsal vagal motor nucleus (DVMN) neurones using an optogenetic approach increases exercise capacity in rats. In heart failure patents, vagus nerve stimulation applied for 15 days was reported to increase the distance of the 6-min walk test. Proof-of-concept studies, primarily in human volunteers, using non-invasive electrical stimulation of either the auricular branch or the cervical bundle of the vagus nerve suggest that maintenance, or augmentation, of vagal activity is feasible, effective and associated with minimal side effects. Although transcutaneous stimulation of auricular nerves is readily accessible, studies lack focus on autonomic activation and have yet to examine effects on exercise capacity.

Here, the investigators describe the protocol for a randomised controlled crossover trial, hypothesizing that bilateral transauricular nerve stimulation (TAN) augments exercise capacity in human volunteers. Furthermore, the investigators aim to identify whether TAN augments exercise capacity in tandem with autonomic changes that are mechanistically implicated in favourably modulating cardiopulmonary fitness.

Recruitment/screening Potential participants (including NHS patients with no specific disease) will be found through posters displayed on NHS premises. After potential participants contact the research team, two independent members of the research team at the clinical research facility shall be involved - one will obtain informed consent while the other will deliver the interventional protocol. The member obtaining consent will call the potential participant and screen them against the eligibility criteria before asking for consent. All eligible participants that undergo screening will be recorded on a screening log on the Investigator Site File, even if they decline the study. Participants will be given a participant information sheet (PIS) one week in advance of the first day of intervention. Written informed consent must be obtained before the first intervention.

Informed consent The principal investigator or suitably qualified nominee will obtain written informed consent from each participant, including provision of a PIS accompanied by the relevant consent form, and an explanation of the aims, methods, anticipated benefits and potential hazards of the trial. All potential participants are free to refuse to enter the trial or to withdraw at any time during the trial, for any reason. If new safety information results in significant changes in the risk/benefit assessment, the PIS and consent form will be reviewed and/or amended accordingly. Participants will be informed that, as defined by the UK Policy Framework for Health and Social Care Research, all documentation will be stored for a minimum of 20 years at the end of the study.

Sample size Consensus CPET guidelines recommend that the VO2peak should be used to assess exercise capacity. The investigators require 28 participants [alpha=0.05; 1-beta=0.9], based on the experimental intervention increasing VO2peak (from each individual's own baseline) by the same degree as high intensity exercise training (which increases VO2peak by 0.51 l·min-1; 95% ci: 0.43 to 0.60 l min-1, SD 0.9). The sample size allows for a dropout rate of 10% per group.

Randomisation Participants are randomly assigned (1:1) by block randomisation to receive active or sham stimulation first to ensure a balance in sample size across groups over time (Power Analysis & Sample Size (PASS) 2021, Utah, USA). Randomisation is performed one week before the first intervention, with a random block size of four. A randomisation sequence is created by a biostatistician who did not participate in the implementation or statistical analysis of trial. Allocation concealment is achieved through sequentially numbered, opaque, sealed envelopes.

Bias/blinding Participants and investigators are blinded to treatment allocations throughout data collection and analysis. Participants and investigators are unable to see the device settings. Participants are instructed by the investigators that the stimulation is imperceptible after determination of the prescription dose. Participants and investigators are also masked to the Holter data, which will be analysed offline by an independent trial statistician not involved with patient recruitment/device application who is masked to the treatment allocations. Interventions are performed at the same time of day to minimise the possible influence of circadian variations.

Data collection Clinical data will be recorded. CPET data will be extracted from the cycle ergometer software (Zan, nSpire). Heart rate data will be analysed using Kubios HRV Premium [version 3.5.0]. Plasma will be stored at -80ºC having been obtained after both intervention periods for exploratory analyses of biomarkers related to autonomic activation. These data will be collected by a member of the research team not involved with administering the interventions, and analysed by an independent member of the research team - both will be masked to the treatment allocations. Data will be entered electronically on a secure database (REDCAP).

Statistical analysis Analyses will be conducted using the intention-to-treat principle, where all participants with a recorded outcome are analysed according to the treatment group to which they were randomised. Baseline participant characteristics will be presented and stratified according to treatment allocation. The primary outcome (absolute change in VO2peak) will be analysed using repeat-measures analysis of variance (intervention allocation x intervention period) (before versus after TAN/sham). For secondary outcomes, heart rate, CPET, HRV data and plasma acetylcholine levels will be compared in each group using repeat-measures analysis of variance. Sensitivity analysis for variables that may affect exercise capacity and/or autonomic measures will also be conducted. The significance level will be set at 0.05. A full statistical analysis plan will be developed prior to analysis and the end of the study.

Trial management/data monitoring The Sponsor organisation is Queen Mary University of London (QMUL). Daily trial management will be coordinated by a trial management group consisting of the Chief Investigator and his/her support staff. An independent study committee will oversee the trial, including assessing the safety of the intervention, reviewing relevant new external evidence, and monitoring the overall conduct of the trial. This committee consists of an independent clinical trialist, lay representative and an independent Chair.

Adverse events Prespecified and any other adverse events directly related to the trial intervention will be recorded.

Confidentiality Information related to participants will be kept confidential and managed in accordance with the Data Protection Act (UK), NHS Caldecott Principles (UK), the Research Governance Framework for Health and Social Care (UK), and the conditions of Research Ethics Committee Approval, or corresponding legislation or approvals for a particular participating country or site. The principal investigator will maintain in strict confidence trial documents (e.g. written consent forms) and confidentiality.

Discussion Exercise capacity serves as an excellent preoperative prognosticator of an individual's ability to cope with the physiological (and pathophysiological) processes underlying ageing. Experimental animal studies and human exercise performance data have shown intact vagal tone enhances exercise capacity. However, acute tissue injury and systemic inflammation disrupt autonomic control. This proof-of-concept study aims to demonstrate the safety, feasibility and efficacy of TAN in augmenting cardiopulmonary fitness in tandem with autonomic changes that are mechanistically associated with favourable modulation of exercise capacity. These healthy volunteer data may offer key insights into potentially accelerating functional rehabilitation.

Experimental data indicate that cardiac vagal activity is a direct determinant of exercise capacity. Persistent autonomic dysfunction directly impairs cardiopulmonary fitness and therefore muscle mass and strength; key determinants of functional recovery cannot be increased. Furthermore, disruption of autonomic-mediated immunoregulatory mechanisms promotes a pro-inflammatory state whereby mechanisms controlling the resolution of inflammation are suppressed. The development and persistence of autonomic dysfunction therefore directly impairs cardiopulmonary fitness and rehabilitation. Therefore, individuals at high risk of morbidity and mortality are characterized by reduced vagal tone and slow heart rate recovery following incremental exercise.

Studies of non-invasive autonomic neuromodulation conducted in healthy volunteers and are susceptible to bias. The investigators utilised a double-blind, open crossover. randomised controlled design to address these issues. Although participants have varying fitness levels before the study, each individual serves as their own control. The use of a designated sham stimulation device is critical to minimise participant and investigator biases. Far more invasive studies have successfully recruited patients into trials where sham procedures served as the key control in cardiac and noncardiac orthopaedic surgery.

Assessing the effects of TAN on exercise capacity in healthy volunteers is broadly generalisable to the general population. Provided that the investigators can confirm in this setting that autonomic changes after TAN occur by measuring HRV, the low cost, non-invasive device used suggests a very low potential risk-to-benefit ratio. Systematic review identified TAN stimulation parameters that alter HRV, although there is no certainty that there may be minimum thresholds for the duration and/or intensity required to be clinically effective. Nonetheless, a 30-minute period of daily tragal stimulation has not been associated with any major adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75y
2. Male or female
3. Able and willing to give informed consent

Exclusion Criteria:

1. Current smoker
2. Currently undertaking a dedicated training/exercise regime (i.e. not sedentary)
3. Excess alcohol intake (as determined via a medical questionnaire)
4. Contraindications to cardiopulmonary exercise testing
5. Pregnancy
6. Auricular dermatitis
7. Unwilling or unable to give consent
8. Inability to understand written and/or verbal English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Change in peak volume of oxygen uptake (VO2peak) | 7 days
  Gold standard measure of exercise capacity

SECONDARY OUTCOMES:
Change in heart rate recovery (HRR) | 7 days
  Gold standard clinical measure of vagal tone. Obtained from exercise bike test.
Change in decline from peak heart rate (PeakHRdecline) after standing from the sitting position | 7 days
  Surrogate marker for HRR. Obtained from orthostatic (sit-to-stand) test.
Change in heart rate variability (HRV) | 7 days
  Time- and frequency-domain components indicative of autonomic balance
Change in plasma acetylcholine levels (PlasmaACh) | 7 days
  Key neurotransmitter of the parasympathetic nervous system; quantified by fluorescence-activated cell sorting

CONTACTS AND LOCATIONS:
Overall Officials: Gareth L Ackland, FRCA, Principal Investigator — Queen Mary University of London
Locations (1):
- William Harvey Research Institute, Barts and The London School of Medicine and Dentistry, Queen Mary University of London, John Vane Science Centre, Charterhouse Square, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
N/A. Double-blinded study. Participants, investigators and analysers masked to data as detailed in study design section.

REFERENCES:
- [Background] Machhada A, Trapp S, Marina N, Stephens RCM, Whittle J, Lythgoe MF, Kasparov S, Ackland GL, Gourine AV. Vagal determinants of exercise capacity. Nat Commun. 2017 May 18;8:15097. doi: 10.1038/ncomms15097. PMID 28516907
- [Background] Gourine AV, Ackland GL. Cardiac Vagus and Exercise. Physiology (Bethesda). 2019 Jan 1;34(1):71-80. doi: 10.1152/physiol.00041.2018. PMID 30540229